CLINICAL TRIAL: NCT02187497
Title: BIBR 277 Capsules Pharmacokinetics Study of Hypertensive Patients
Brief Title: Pharmacokinetics of BIBR 277 in Hypertensive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.268
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

ARMS (3):
- Low dose of BIBR 277 (Experimental)
  Interventions: Drug: Low dose of BIBR 277
- Medium dose of BIBR 277 (Experimental)
  Interventions: Drug: Medium dose of BIBR 277
- High dose of BIBR 277 (Experimental)
  Interventions: Drug: High dose of BIBR 277

INTERVENTIONS:
Drug: Low dose of BIBR 277
  Arms: Low dose of BIBR 277
Drug: Medium dose of BIBR 277
  Arms: Medium dose of BIBR 277
Drug: High dose of BIBR 277
  Arms: High dose of BIBR 277

SUMMARY:
The pharmacokinetic profile of BIBR 277 single dose given in capsule form to hypertensives was evaluated. The results of the present study are to be used in the Japanese population pharmacokinetics analysis

ELIGIBILITY:
Inclusion Criteria:

* Age: >=20 years
* Sex: Either male or female
* Patient status: Either inpatient or outpatient, provided that the patient was available for hospitalisation from the day before the trial medication administration until the morning of the day after administration
* BP: Sitting systolic and diastolic blood pressures (SBP and DBP) taken the day before administration should be >= 150 mmHg and >= 90 mmHg, respectively. Patients undergoing treatment with other antihypertensives were not excluded provided the above criteria were satisfied.

Exclusion Criteria:

* Malignant hypertension
* Renovascular hypertension
* Severe heart failure (NYHA functional class III - IV), unstable angina pectoris, or history of myocardial infarction (within 6 months of onset)
* Atrioventricular conduction disturbance (degree II to III), atrial fibrillation, or serious arrhythmia
* Symptoms of cerebrovascular disorder
* Serious hepatic dysfunction
* Renal function disorder (serum creatinine >= 4.0 mg/dL)
* Known hypersensitivity to angiotensin II receptor antagonists
* Hyperkalaemia (potassium >= 5.5 milliequivalents per liter (mEq/L))
* Treatment with the other investigational drug within 6 months of initiation of the present study
* Pregnant, breast feeding, possibly pregnant or planning to become pregnant during this study
* Previous treatment with the trial medication of the present study
* Otherwise judged ineligible by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 1998-06; Primary Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BIBR 277 in plasma from 0 to 24 hours (AUC0-24hr) | Pre-dose up to 24 hours after start of treatment
Mean residence time of BIBR 277 in the body from 0 to 24 hours (MRT0-24hr) | Pre-dose up to 24 hours after start of treatment
Maximum measured concentration of BIBR 277 in plasma (Cmax) | Pre-dose up to 24 hours after start of treatment
Time from dosing to the maximum concentration of BIBR 277 in plasma (tmax) | Pre-dose up to 24 hours after start of treatment
Terminal elimination half-time of BIBR 277 in plasma (t1/2) | Pre-dose up to 24 hours after start of treatment

SECONDARY OUTCOMES:
Changes from baseline in blood pressure (systolic, diastolic, and mean) | Pre-dose up to 14 days after start of treatment
Changes from baseline in pulse rate | Pre-dose up to 14 days after start of treatment
Number of patients with adverse events | Up to 29 days
Changes from baseline in laboratory test values | Pre-dose up to 14 days after start of treatment